CLINICAL TRIAL: NCT03433209
Title: Electrosurgery Wars;Ligasure or Enseal in Total Laparoscopic Hysterectomy: A Randomised Controlled Trial
Brief Title: Electrosurgery Wars;Ligasure or Enseal in Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Karadag, MD, Associate Professor, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9-1
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Task Performance
Keywords: Advanced bipolar energy devices; ENSEAL; LigaSure; Operative time; Total laparoscopic hysterectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ligasure device (Active Comparator): This group of women undergoing hysterectomy were randomized to the Ligasure energy device
  Interventions: Device: Ligasure device
- Articulating Enseal (Active Comparator): This group of women undergoing hysterectomy were randomized to the articulating Enseal energy device
  Interventions: Device: Articulating Enseal

INTERVENTIONS:
Device: Ligasure device — Vessel-sealing device used for laparoscopic hysterectomy
  Arms: Ligasure device
Device: Articulating Enseal — Vessel-sealing device used for laparoscopic hysterectomy
  Arms: Articulating Enseal

SUMMARY:
The effect of two different bipolar instruments were compared in terms of operative time, total operative time, intra-operative blood loss and intra-operative and postoperative complications. Devices included the LigaSure™ Maryland Jaw 5 mm laparoscopic instrument (LigaSure; LF 1737, Covidien, Mansfield, MA, USA) and ENSEAL™ G2 Articulating Straight 5mm Tissue Sealer (ENSEAL; NSLG2S35A, Ethicon Endo-surgery, US, LLC).

DETAILED DESCRIPTION:
This study is a single-center, single-blinded, randomized control trial that was conducted at the University of Health Sciences Antalya Training and Research Hospital.

The study was single-blinded in that the patient was not informed of their group assignment; it is impossible to blind the surgeon using the devices.

Methods and Procedures:

Patients were recruited from outpatient clinics and informed about the study before enrollment. Women aged over 18 years scheduled for laparoscopic hysterectomy for benign indications between June 2016 and November 2017 were included in the study after obtaining written consent.

Women who had given consent were randomized one day before surgery to one of two groups:

Group 1: The Ligasure device used during the hysterectomy. Group 2: The articulating Enseal device used during the hysterectomy.

Inclusion Criteria:

* Age 18 or older
* Able and willing to provide informed consent

Exclusion Criteria:

* Under 18 years of age
* Suspected malignancy

Surgical technique:

All laparoscopic procedures were performed under general anesthesia. An experienced surgeon, who has an experience of over 100 cases of TLH with both LigaSure and Enseal, performed all the procedures. Because both devices have long been used in the operations, they are always ready for use in our operation rooms. During the study, the first assistant was always a second or a third year assistant surgeon and the second assistant holding the uterine manipulator was a first year assistant surgeon. Operative time was recorded in minutes with a digital watch by a first year resident by dictation of the primary surgeon of the start and stop times.

After positioning the patient in lithotomy position and placement of a Foley catheter, a Rumi II (CooperSurgical, Inc, Trumbull, CT, USA) uterine manipulator with Koh cup (Bard Medical, Covington, GA, USA) of appropriate size was placed. The first assistant stood on the right side of the patient and held the camera. The second assistant held the uterine manipulator. The abdominal cavity was entered by direct trocar insertion. The site of insertion varied, being the umbilicus or Lee-Huang point, according to the size of the uterus. After pneumoperitoneum was obtained, the patient was positioned in the Trendelenburg position and three additional trocars, all 5 mm in size, were inserted from both inguinal regions and suprapubic region. Following exploration of the abdominal cavity, adhesiolysis was performed where necessary. The round ligaments were sealed and transected, the bladder peritoneum was opened, the utero-ovarian ligaments were sealed and cut, the bladder peritoneum was dissected from the vagina, the uterine vessels were skeletonized, sealed and dissected followed by sacro-uterine ligament dissection and finally the vaginal wall on the rim of the vaginal part of the uterine manipulator was cut by Harmonic AceTM. The uterus was removed vaginally in all operations but in case of large uteri, either a Chardonnen's morcellation knife (Karl Storz GmBH, Tuttlingen, Germany) or a power morcellator was used for uterine section before retrieval. The vaginal cuff was closed by laparoscopic stitching with number 1 Vicryl suture. In cases where bilateral or unilateral salpingo-oophorectomy was also indicated, the procedure was performed after removal of the uterus in order to prevent interference with operative time which was our primary outcome measure. To seal and transect uterine attachments, the LigaSure™ Maryland Jaw 5 mm laparoscopic instrument (LigaSure; LF 1737, Covidien, Mansfield, MA, USA), using the ForceTriadTM Energy Platform (Covidien, Boulder, CO, USA) was used in one group and ENSEAL™ G2 Articulating Straight 5mm Tissue Sealer (ENSEAL; NSLG2S35A, Ethicon Endo-surgery, US, LLC) using the Ethicon GEN11TM generator (Ethicon Endo-surgery, US, LLC) was used in the other group.

Follow-up was performed on postoperative day 7, and then at 1 month.Patients were also seen at our clinic if they developed symptoms between follow-up visits and complications recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able and willing to provide informed consent
* Undergoing total laparoscopic hysterectomy

Exclusion Criteria:

* Under 18 years of age
* Suspected malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Operative time | 16 months
  Defined as time from start of sealing and transection of the round ligament until start of colpotomy, was the primary endpoint.

SECONDARY OUTCOMES:
Total operative time | 16 months
  Time from placement of the first trocar until removal of all trocars
Intra-operative estimated blood loss | 16 months
  Calculated by subtracting total volume of irrigated fluid from the amount measured in the aspiration bag after positioning the patient in reverse Trendelenburg position at the end of the operation
Intra-operative complications | 16 months
  Visceral or vascular injury, hemorrhage, conversion to laparotomy, mechanical or functional device failure